CLINICAL TRIAL: NCT02397005
Title: Randomized, Double-blind, Placebo-controlled Study of the Tolerability and Pharmacokinetics of Ascending Single and 14-day Repeated Oral Doses of ZL-2102 With a Pilot Investigation of Food Effect in Healthy Male Subjects
Brief Title: Study of the Tolerability and Pharmacokinetic of ZL-2102 With an Investigation of Food Effect in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zai Lab Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZL-2102-SAD/FED/MAD
Record Dates: First submitted 2015-02-27; First posted 2015-03-24 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZL-2102 (Active Comparator): Planned to be administrated in an ascending manner: 5,20,60,150,300,500,750mg
  Interventions: Drug: ZL-2102
- Placebo (Placebo Comparator): Placebo matching ZL-2102
  Interventions: Drug: Placebo matching ZL-2102

INTERVENTIONS:
Drug: ZL-2102 — A selective and reversible inhibitor of Hematopoietic Prostaglandin D Synthase (HPGDS).
  Arms: ZL-2102
Drug: Placebo matching ZL-2102
  Arms: Placebo

SUMMARY:
The first-in-man study are designed as below to assess safety, tolerability, and preliminary pharmacokinetics of ZL-2102.

* Double-blind randomized, placebo-controlled ascending single oral doses (Part 1, ZL-2102-SAD);
* Open-label, randomized, 2-sequence, 2-period, 2-treatment crossover (Part 2, ZL-2102-FED);
* Double-blind randomized, placebo-controlled, ascending repeated oral doses for 14 days (Part 3, ZL-2102-MAD).

A total of 104 subjects will be enrolled.

DETAILED DESCRIPTION:
There are 3 parts to the study. Subjects will be randomized to receive ZL-2102 or matching placebo (3: 1 ratio) in Parts 1 and Part 3 of the study. Subjects in Part 2 will be randomized 1:1 to receive ZL-2102 in each possible treatment sequence (fed/fasted or fasted/fed).

In Part 1 (ZL-2102-SAD), the safety, tolerability and pharmacokinetics of the study drug or placebo will be tested after a single dose in the form of a capsule when given after an overnight fast. There will be 7 groups. Groups 1 to 7 will have a total of 8 participants in each group, with 56 participants total in all 7 groups. Each group will receive a different dose of the study drug or placebo in the following order of strength: 5, 20, 60, 150, 300, 500, 750 mg. Plasma samples will be collected in 0H,0H30M,1H,2H,3H,4H,5H,6H,8H,10H,12H,16H,24H,48H and on Day 8. Urine samples will be collected at 0-4,4-8,8-12,12-24,24-28H intervals. Subjects will be confined to the unit for 3 days and the follow-up observation period is 7 days after the administration.

Part 2 of the study (ZL-2102-FED) will test the effect of a high-fat meal on safety, tolerability and pharmacokinetics of the study drug after a single dose in 12 healthy male subjects. Choice of dose of ZL-2102 will be made based on review of the blinded preliminary safety, tolerability and pharmacokinetics data in Part 1. No subjects will receive placebo in Part 2. Two single doses separated by at least a 7-day wash-out period. One dose will be given under fed (standardized high-fat breakfast) and one will be under fasted conditions.

Part 3 of the study (ZL-2102-MAD) will test the safety, tolerability and pharmacokinetics of the study drug after repeated doses of the study drug. Three dose level groups (9 active and 3 placebo) with 12 healthy male subjects will be enrolled.Choice of the actual daily ZL-2102 doses will be made based upon a review of the blinded preliminary safety, tolerability, and pharmacokinetics data in Part 1. Three ascending once-daily repeated doses of ZL-2102 or placebo for 14 days or, alternatively, twice daily for 14 days if indicated by pharmacokinetics parameters from Part 1 (ZL-2102-SAD). If the dose needs to be twice daily, the total daily doses will be given half in the morning and half in the evening 12 hours later. Dose will be administered either under fed or fasted conditions depending on blinded Part 2 (ZL-2102-FED) results.

The trial will be conducted in Linear Clinical Research Ltd.by Principle Investigator Janakan Krishnarajah,MD and his team.

ELIGIBILITY:
Inclusion Criteria:

* Male subject, between 18 and 45 years of age inclusive.
* Body weight between 50.0 and 100.0 kg inclusive, body mass index (BMI) between 18.0 and 30.0 kg/m² inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 5 minutes resting in a semi recumbent position.
* Normal standard 12-lead ECG after 5 minutes resting in a semi recumbent position.
* Laboratory parameters within the normal range, or considered not clinically significant by the Investigator.
* Subject returns a negative result to the Serology,Urine drug screen and alcohol breath tests.
* Having given written informed consent prior to any procedure related to the study.
* Not under any administrative or legal supervision.
* Males must agree to use adequate contraception for the duration of the study and for 3 months post completion of dosing.
* Subject agrees to the following study restrictions:

  1. Subject will not consume citrus fruits and their juices for 5 days before the start of the study, and for the duration of the study.
  2. Subject will not consume alcohol, tea, coffee, chocolate, quinine or caffeine-containing beverages from Day 1 and for the duration of the study.
  3. Subject will note smoke or use tobacco from Day 1 and for the duration of the study.
  4. Subject will avoid intensive physical activity from Day 1 and for the duration of the study.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteo-muscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months prior to Screening.
* Symptomatic postural hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension defined by a decrease in systolic blood pressure ≥ 20 mmHg within 3 minutes when changing from the supine to the standing position.
* Presence or history of drug hypersensitivity, or allergic disease (excluding hay fever) diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption >40 grams per day).
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Excessive consumption of beverages with xanthine bases (>4 cups or glasses per day).
* Any prescription medication within 14 days and any over the counter medication within 7 days before Screening or within 5 times the elimination half-life or Pharmacodynamic half-life of that drug whichever is longest unless approved by both the Investigator and the Medical Monitor; any vaccination within the last 28 days. If necessary, paracetamol (acetaminophen) may be administered with the approval of the Investigator.
* Any subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Receipt of any investigational study drug within 30 days prior to screening.
* Any subject who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in the conduct of the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Part1,ZL-2102-SAD: Safety as measured by Adverse Events | 8 days
Part2,ZL-2102-FED: Safety as measured by Adverse Events | 15 days
Part3,ZL-2102-MAD: Safety as measured by Adverse Events | 21 days
Peak Plasma Concentration (Cmax) of ZL-2102 | 48 hours
Area under the plasma concentration versus time curve (AUC) of ZL-2102 | 48 hours

SECONDARY OUTCOMES:
Part1,ZL-2102-SAD: Safety as measured by Physical examination, body weight, hematology, biochemistry, urinalysis, vital signs and 12-lead ECG. | 8 days
Part2,ZL-2102-FED: Safety as measured by Physical examination, body weight, hematology, biochemistry, urinalysis, vital signs and 12-lead ECG. | 15 days
Part3,ZL-2102-MAD: Safety as measured by Physical examination, body weight, hematology, biochemistry, urinalysis, vital signs and 12-lead ECG. | 21 days

OTHER OUTCOMES:
Peak Urine Concentration (Cmax) of ZL-2102 | 48 hours
Area under the urine concentration versus time curve (AUC) of ZL-2102 | 48 hours
Part3,ZL-2102-MAD: Concentration of 2,3-dinor-6-keto-PGF1α as Prostaglandin I2 metabolite in urine. | 48 hours
Part3,ZL-2102-MAD: Concentration of 13,14-dihydro-15-keto PGA2 and 13,14-dihydro-15-keto PGE2 as Prostaglandin E2 metabolite in urine. | 48 hours
Part3,ZL-2102-MAD: Concentration of 11-dehydrothromboxane B2 as Thromboxane A2 metabolite in urine. | 48 hours
Part3,ZL-2102-MAD: Concentration of 13, 14-dihydro-15-keto PGF2a as Prostaglandin F2α in plasma. | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Unit, Perth, Australia